CLINICAL TRIAL: NCT06712771
Title: A Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of VSA003 Injection in Chinese Adolescents and Adults with Homozygous Familial Hypercholesterolaemia (HoFH)
Brief Title: A Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of VSA003 in Chinese HoFH Patients
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Visirna Therapeutics HK Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VSA003-3001
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Homozygous Familial Hypercholesterolemia (HoFH)
MeSH Terms: conditions — Homozygous Familial Hypercholesterolemia | interventions — zodasiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VSA003 (Experimental): subcutaneous injections
  Interventions: Drug: VSA003
- Placebo (Placebo Comparator): subcutaneous injections
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VSA003 — subcutaneous injections
  Other Names: AROANG3; Zodasiran
  Arms: VSA003
Drug: Placebo — subcutaneous injections
  Arms: Placebo

SUMMARY:
Significant reduction in ANGPLT3 levels is expected to reduce plasma LDL-C and TG levels and may lead to the reduction of risk of coronary heart disease and cardiovascular events associated with hypertriglyceridemia and LDL-C in subjects with persistent dyslipidemia. In this clinical study, the efficacy and safety of VSA003, an RNAi-based therapeutic targeting ANGPTL3, will be evaluated in subjects with HoFH.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged ≥ 12 years and weighing ≥ 40 kg at the time of ICF signature;
* Patients with HoFH who meet genetic or clinical diagnosis;
* Willing to follow a daily low-fat diet for the duration of the study;
* Receiving stable and tolerable lipid-lowering therapy prior to LDL-C testing during the screening period;
* Fasting LDL-C ≥ 2.6 mmol/L.

Exclusion Criteria:

* Have received or are receiving targeted ANGPTL3 treatment within 5 months or 5 half-lives, whichever is longer, prior to screening;
* Fasting TG ≥ 4.5 mmol/L at screening;
* Presence of uncontrolled endocrine disease affecting lipids or lipoproteins;
* Weight change of more than 10% in the 4 weeks prior to randomisation;
* Initiation of a new dietary plan or significant differences from previous dietary structure and habits within 4 weeks prior to screening;
* Women who are pregnant (including planned pregnancies) or breastfeeding;
* Refusal to limit alcohol consumption to moderate limits and below during the study period, specifically no more than 14 units per week;
* Uncontrolled hypertension (blood pressure > 160/100 mmHg at screening);
* New York Heart Association (NYHA) class IV heart failure or left ventricular ejection fraction <30% within 12 months prior to screening;
* History of major surgery within 12 weeks prior to baseline, or planning to undergo major surgery during the study;
* Known allergy to any component of the study drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in serum LDL-C at month 6 | At month 6

SECONDARY OUTCOMES:
Percent change and absolute change in serum ANGPTL3 levels from baseline at month 6 | At month 6
Percent change and absolute change in serum LDL-C, ApoB, non-HDL-C, VLDL-C, TC and TG levels from baseline | Up to month 6, Up to month 18
Percent change and absolute change in serum HDL-C, ApoC-III, ApoC-II, ApoA-I, ApoA-V and Lp[a] levels from baseline | Up to month 6, Up to month 18
Percentage of patients achieving ≥30% reduction in serum LDL-C from baseline | At month 6, At month 18
Percentage of patients achieving ≥50% reduction in serum LDL-C from baseline | At month 6, At month 18
Number of Participants with Adverse Events | Up to month 6, Up to month 18
Number of Participants with Anti-Drug Antibodies (ADAs) to VSA003 Over Time | Up to month 6, Up to month 18
Correlation between VSA003 serum concentrations and QT intervals | Up to month 6, Up to month 18

IPD SHARING:
Plan to Share IPD: No